CLINICAL TRIAL: NCT04154696
Title: APHP Plateform for Assessement of Hepatic Grafts Initialy Discarded by Normothermic Perfusion
Brief Title: APHP Plateform of Normothermic Perfusion for Rehabilitation of Hepatic Grafts
Acronym: PENOFOR
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P170605J
Record Dates: First submitted 2019-08-21; First posted 2019-11-06 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-08

CONDITIONS: Liver Diseases
Keywords: Steatotic liver graft; Liver transplantation; Normothermic perfusion
MeSH Terms: conditions — Liver Diseases

STUDY DESIGN:
Intervention Model Description: Liver transplantation of a graft after assessment by normothermic perfusion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Normothermic perfusion of a graft (Experimental)
  Interventions: Procedure: Liver transplantation of a graft after assessment by normothermic perfusion

INTERVENTIONS:
Procedure: Liver transplantation of a graft after assessment by normothermic perfusion — Liver transplantation of a graft after assessment by normothermic perfusion

SUMMARY:
This study aimed to evaluate fatty liver grafts, considered as unsuitable for upfront liver transplantation, by using normothermic perfusion. Grafts have to be allocated to one of 3 liver transplantation centres of Paris. After evidence of viability while on perfusion, these grafts will be transplanted to recipients with an estimated waiting time > 6 months.

DETAILED DESCRIPTION:
In this study, the coordinator investigator proposes to build a platform for perfusing in normothermic conditions all grafts with histologically proven macrosteatosis ≥ 30% that will be considered as unsuitable for upfront LT. These grafts have to be alloacted to one of the 3 liver transplantation centers of Assistance Publique des Hôpitaux de Paris. Eligible grafts (macrosteatosis ≥ 30%, no severe fibrosis or cirrhosis) will be shipped to the platform for normothermic perfusion. Perfusion will be started provided that cold ischemia time do not exceed 8 hours. Parameters of grafts viability (lactates, bile production, flow) will be monitored. After a minimum of 4 hours of normothermic perfusion (not exceeding 16 hours), grafts fulfilling strict criteria (homogeneous aspect of the liver without any necrotic regions, lactates < 2.5 mmol/l and continuous production of bile with at least one of the following criteria: pH of perfusate > 7.3, arterial flow > 150 ml/min and portal flow > 500 ml/min, homogeneous perfusion of the graft) will be considered suitable for transplantation. Recipient will be transferred to the operating room, and first phase of LT (i.e, laparotomy and total hepatectomy) will be started. Simultaneously, grafts will be shipped to the center of initial allocation. Perfusion will be pursued during the transport from the platform to the recipient. Recipients (≥18 years and ≤ 70 years) have to be enlisted for LT with an estimated waiting time > 6 months (i.e., MELD score < 25) and who signed an informed consent.

ELIGIBILITY:
Inclusion Criteria:

* patients enlisted for liver transplantation for liver disease or HCC (AFP score≤ 2);
* Ongoing cotraception in women of reproductive age ;
* Patient with social security ;
* informed signed consent

Exclusion criteria:

* Extra-hepatic tumor disease;
* Re-transplantation ;
* Pregnancy or brest-feeding;
* Patients participting in another study;
* Patients under psychiatric treatment;
* Patients under tutorship or curatorship

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2019-10-28 (Estimated); Primary Completion 2021-07-01 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
To determine the proportion of grafts that can be transplanted after evaluation by normothermic perfusion (Hypothesis 50%) with a 3-year graft survival ≥ 90% | 3 months
  Graft survival

SECONDARY OUTCOMES:
Proportion of hepatic grafts allocated to the 3 transplant centres of Paris and considered as initially not transplantable during the study period | 36 months
  Proportion of hepatic grafts allocated to the 3 transplant centres of Paris and considered as initially not transplantable during the study period
Proportion of fatty grafts allocated to the 3 transplant centres of Paris and considered as initially not transplantable during the study period eligible for normothermic perfusion | 36 months
  Proportion of fatty grafts allocated to the 3 transplant centres of Paris and considered as initially not transplantable during the study period eligible for normothermic perfusion
Proportion of grafts perfused | 36 months
  Proportion of grafts perfused
Proportion of grafts that were transplanted after perfusion | 36 months
  Proportion of grafts that were transplanted after perfusion
Time interval until liver function recovery while on normothermic perfusion (according to viability criteria defined above) | 15 hours
  Time interval until liver function recovery while on normothermic perfusion (according to viability criteria defined above)
Proportions of grafts transplanted after normotheric perfusion wthout early allograft dysfunction (according to Olthoff definition) | one month
  Proportions of grafts transplanted after normotheric perfusion wthout early allograft dysfunction (according to Olthoff definition)
Time interval until liver function recovery after transplantation | one day
  Time interval until liver function recovery after transplantation
One-month overall survival (without retransplantation or graft dysfunction) | one month
  One-month overall survival (without retransplantation or graft dysfunction)
One -year graft survival | one year
  One -year graft survival
Comparison of 3-months graft survival with a control group of graft considered as initially transplantable | 3 months
  Comparison of 3-months graft survival with a control group of graft considered as initially transplantable
Waiting time between the two groups | 36 months
Incidence of biliary stenosis (anastomotic or non anastomotic) defined by cholangio MRI at one year | 12 months
  Incidence of biliary stenosis (anastomotic or non anastomotic) defined by cholangio MRI at one year

CONTACTS AND LOCATIONS:
Locations (1):
- AP-HP, Paul Brousse Hospital, Villejuif, France

IPD SHARING:
Plan to Share IPD: Undecided